CLINICAL TRIAL: NCT00487292
Title: The Effects of a Combination of Napping and Bright Light Pulses on Shift Workers Sleepiness at the Wheel A Pilot Study
Brief Title: Naps and Pulses of Bright Light in Shift Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HDCSRE-003
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2007-06

CONDITIONS: Sleep
Keywords: accidents; shift work; sleepiness; naps; bright light pulses; sleep
MeSH Terms: conditions — Sleepiness | interventions — N-(4-aminophenethyl)spiroperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: naps and pulses of bright light

SUMMARY:
Design: paired trials without and with naps and bright light. Setting: Real driving on a private road circuit. Environmental controlled car. Participants: 9 shift workers on tree shifts (morning-afternoon-night) Measurements: Sleepiness at the wheel was measured by ambulatory polysomnography and assessed using 30 seconds segments of recordings when the percentage of theta EEG was at least 50% (15 seconds) of the period recorded. Subjects were also called to rate their sleepiness on the 7-point Stanford Sleepiness Scale (SSS).

Intervention: Participants drove the same car on two similar 24 hours periods of work, with three pilots in each shift (morning, afternoon, night), separated by three weeks. During the baseline period, the subjects were told to manage their rest as they usually do in the real life. During the second experimental period, they had to rest lied in a dark room during two naps of 20 minutes and then exposed to bright light pulse (5000 lux) during 10 minutes.

DETAILED DESCRIPTION:
Results are submitted to publication

ELIGIBILITY:
Inclusion Criteria:

* A professional experience of at least one year

Exclusion Criteria:

* With an history of chronic disease,treatments (or toxic)
* Subjects with a suspicion of sleep disorders
* Snorers

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2003-04; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
EEG sleepiness at the wheel | two periods of 8 hours driving

SECONDARY OUTCOMES:
subjective sleepiness at the stanford sleepinesss scale | two periods of 8 hours driving

CONTACTS AND LOCATIONS:
Overall Officials: damien leger, M.D, Ph.D, Principal Investigator — Centre du Sommeil Hotel Dieu; pierre philip, M.D, Ph.D, Study Director — Hopital Pellegrin Bordeaux
Locations (1):
- Centre du Sommeil Hôtel Dieu de Paris, 1 place Parvis Notre Dame, Paris, France

REFERENCES:
- [Background] Leger D, Annesi-Maesano I, Carat F, Rugina M, Chanal I, Pribil C, El Hasnaoui A, Bousquet J. Allergic rhinitis and its consequences on quality of sleep: An unexplored area. Arch Intern Med. 2006 Sep 18;166(16):1744-8. doi: 10.1001/archinte.166.16.1744. PMID 16983053
- [Background] Philip P, Taillard J, Moore N, Delord S, Valtat C, Sagaspe P, Bioulac B. The effects of coffee and napping on nighttime highway driving: a randomized trial. Ann Intern Med. 2006 Jun 6;144(11):785-91. doi: 10.7326/0003-4819-144-11-200606060-00004. PMID 16754920